CLINICAL TRIAL: NCT04844346
Title: The Effect of Plant Stanol Ester Consumption on the Vaccination Response to a COVID-19 Vaccine
Brief Title: Plant Stanol Esters and COVID-19 Vaccination Response
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was dependent on finding participants that had to receive an initial COVID-19 vaccination and we were unable to find new participants anymore.
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Raisio Nutrition Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: METC 21-013
Record Dates: First submitted 2021-04-13; First posted 2021-04-14 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Overweight and Obesity
Keywords: Overweight; Obesity; COVID-19 vaccine; Immune system; Vaccination response
MeSH Terms: conditions — Overweight; Obesity | interventions — COVID-19 Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plant stanol group (Experimental): This arm receives 4g of plant stanols per day (delivered as plant stanol esters) by consuming mini drinks (100 mL each).
  Interventions: Dietary Supplement: Plant stanol mini drinks; Biological: COVID-19 vaccine
- Placebo group (Placebo Comparator): This arm receives mini drinks without added plant stanols (delivered as plant stanol esters).
  Interventions: Dietary Supplement: Placebo mini drinks; Biological: COVID-19 vaccine

INTERVENTIONS:
Dietary Supplement: Plant stanol mini drinks — Oat milk based mini drinks (100 mL) containing 2g plant stanols each (delivered as plant stanol esters).
  Arms: Plant stanol group
Dietary Supplement: Placebo mini drinks — Oat milk based mini drinks (100 mL) without added plant stanols (delivered as plant stanol esters).
  Arms: Placebo group
Biological: COVID-19 vaccine — First dose of one of the COVID-19 vaccines. Participants have to wait until they are invited to receive the vaccine by the government; this study does not interfere with national planning of the vaccines.

SUMMARY:
Plant stanols are known to lower low-density lipoprotein cholesterol (LDL-C). However, studies have suggested that these compounds also beneficially influence the immune system, e.g. increasing vaccine-specific antibody titers. BMI has previously been negatively associated to vaccination responses. If plant stanols indeed have beneficial effect on the immune system, people with overweight or obesity might benefit from consuming plant stanols prior to receiving the COVID-19 vaccination. The primary objective of this study is to demonstrate clinical benefits of consumption of plant stanols (delivered via products enriched with plant stanol esters) on the vaccination response to a COVID-19 vaccine in overweight or obese patients. The main study endpoint is vaccination response to a COVID-19 vaccine. Secondary endpoints include amongst others hematological, inflammatory and immunological parameters (e.g. hs-CRP, leukocyte differential count) and metabolic markers (e.g. blood lipid profiles, plasma glucose, serum insulin, HOMA-IR).

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Aged 18 years or older
* BMI between 27 and 35 kg/m2
* Currently not using products containing plant sterols or stanols (products with a cholesterol lowering claim of Becel ProActiv, Benecol, Danacol, store brands)
* Willing to abstain from products containing plant sterols or stanols during the study (products with a cholesterol lowering claim of Becel ProActiv, Benecol, Danacol, store brands)
* Willing to keep the intake of fish oil and vitamin supplements constant

Exclusion Criteria:

* Already received COVID-19 vaccination
* Already had a positive test for COVID-19 (this includes all types of tests, e.g. PCR tests or antibody tests)
* Allergy to an ingredient of the mini drinks
* Having donated blood within one month prior to the start of the study, or planning to donate blood during the study
* Pregnant women
* Breastfeeding women
* Excessive alcohol use (>20 consumptions per week)
* Regular use of soft or hard drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Vaccine specific antibody titers | Change T=0 and T= 4 weeks
  The response to the COVID-19 vaccine will be measured by quantifying specific antibody titers (vaccine specific IgG and IgM). These titers will be measured in blood samples collected weekly during the month after vaccination by suitable ELISAs.

SECONDARY OUTCOMES:
Immune parameters (1) | T=-1 (start study), T=0 (day before vaccination), T=4 weeks after vaccination
  Cytokine production by PBMCs after stimulation with antiCD3-antiCD28 antiCD28 antibodies using the TruCulture system
Immune parameters (2) | T=-1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  hsCRP
Leukocyte count | T=-1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  Number of leukocytes measured in EDTA plasma
Leukocyte differential count | T=-1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  Number of subgroups of leukocytes measured in EDTA plasma
Fasted metabolism (1) | T=-1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  Serum non-cholesterol sterols and stanols
Fasted metabolism (2) | T=-1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  Serum lipid and lipoprotein profile
Fasted metabolism (3) | T=-1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  Glucose metabolism (including e.g. plasma glucose, serum insulin and calculated HOMA-IR)
Anthropometry (1) | T=-1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  Body weight
Anthropometry (2) | T=-1 (start study)
  Height
Anthropometry (3) | T=-1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  Waist circumference
Anthropometry (4) | T=-1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  Hip circumference
Anthropometry (5) | T=-1 (start study), T=0 (day before vaccination), weekly in the month after vaccination (T1-T4)
  Waist-to-hip ratio
Diet | T=-1 (start study) and T=4 weeks after vaccination (end study)
  Food frequency questionnaire is used to determine if the participants maintain their habitual diet and to determine if the participants do not consume plant stanols and/or sterols outside the intervention
Diary outcomes (1) | T=-1 (start study) until T=4 weeks after vaccination (end of study)
  General illness
Diary outcomes (2) | T=0 (day before vaccination) until T=4 weeks after vaccination (end of study)
  Side effects COVID-19 vaccine
Diary outcomes (3) | T=-1 (start study) until T=4 weeks after vaccination (end of study)
  Medication intake

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum Plat, PhD, Principal Investigator — Maastricht University Medical Center; Ronald P Mensink, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] van Brakel L, Mensink RP, Lutjohann D, Plat J. Plant stanol consumption increases anti-COVID-19 antibody responses, independent of changes in serum cholesterol concentrations: a randomized controlled trial. Am J Clin Nutr. 2024 Apr;119(4):969-980. doi: 10.1016/j.ajcnut.2024.01.017. Epub 2024 Jan 24. PMID 38278364